CLINICAL TRIAL: NCT01610895
Title: A Randomized Prospective Trial Comparing Split Dose Polyethylene Glycol-Based Lavage With Clear Fluids Versus Split Dose Polyethylene Glycol-Based Lavage With a Low-Residue Diet in Preparation of Patients for Colonoscopy.
Brief Title: Split Dose Polyethylene Glycol (PEG) + Clear Fluids Versus Split Dose PEG + Low-Residue Diet
Acronym: BP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Alaa Rostom, Associate Professor - Medical Director, Colon Cancer Screening Centre, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 24206
Record Dates: First submitted 2012-05-30; First posted 2012-06-04 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-05

CONDITIONS: Colorectal Cancer
Keywords: Colonoscopy; low fibre diet; clear fluids; Bowel Preparation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Split-dose PEG Based Lavage (2L + 2L) + Low-fiber Diet (Active Comparator): Patients randomized to this arm will have a split-dose Polyethylene Glycol Based lavage (2L + 2L), have a low-fibre diet 4 days prior to Colonoscopy and the day before Colonoscopy, have a low-fibre breakfast, a low-fibre lunch by 2PM and then drink only clear fluids until after the procedure is completed.
  Interventions: Other: Split-dose PEG Based Lavage (2L + 2L) with Low-Fibre Lunch Dietary instructions
- Split-dose PEG Based Lavage (2L + 2L) + Clear fluid diet (Placebo Comparator): Patients randomized to this arm will have a split-dose Polyethylene Glycol Based lavage (2L + 2L), have a low-fibre diet 4 days prior to Colonoscopy and the day before Colonoscopy, have a low-fibre breakfast and then drink only clear fluids until after the procedure is completed.
  Interventions: Other: Split-dose PEG Based Lavage (2L + 2L) with Standard Dietary Instructions

INTERVENTIONS:
Other: Split-dose PEG Based Lavage (2L + 2L) with Low-Fibre Lunch Dietary instructions — Patients will be instructed to arrive for colonoscopy at or after 10 AM. Preparation Instructions: At 8pm the day before the colonoscopy drink 2L of PEG within 2 hours. Starting 5 hours before their arrival time on the day of Colonoscopy, drink the remaining 2L of PEG within 2 hours.
  Dietary Instructions: Low fibre diet for 4 days prior to Colonoscopy. The day before Colonoscopy, low-fibre breakfast, a low-fibre lunch by 2 PM (Created from the table of acceptable foods) and then drink clear fluids until after the procedure is completed.
  Arms: Split-dose PEG Based Lavage (2L + 2L) + Low-fiber Diet
Other: Split-dose PEG Based Lavage (2L + 2L) with Standard Dietary Instructions — Patients will be instructed to arrive for colonoscopy at or after 10 AM.
  Preparation Instructions: At 8pm the day before the colonoscopy drink 2L of PEG within 2 hours. Starting 5 hours before their arrival time on the day of Colonoscopy, drink the remaining 2L of PEG within 2 hours.
  Dietary Instructions: Low fibre diet for 4 days prior to Colonoscopy. The day before Colonoscopy, low-fibre breakfast and then drink clear fluids until after the procedure is completed.
  Arms: Split-dose PEG Based Lavage (2L + 2L) + Clear fluid diet

SUMMARY:
The objective of the study is to examine the effect of adding a strict low-residue lunch on the day before colonoscopy has on clinical efficacy and patient tolerability of bowel preparation, with patients receiving split-dose Polyethylene Glycol Based Lavage.

The primary outcomes will be 1) quality of preparation in cleansing the colon and 2) patient satisfaction

DETAILED DESCRIPTION:
All patients between the ages 18-74 years referred to the Forzani MacPhail Colon Cancer Screening Centre (CCSC) in Calgary, Alberta, Canada for colonoscopy will be considered for inclusion. During pre-assessments at the clinic, patients are asked to consider a general research consent. If they agree to that, then they will be approached for consideration of participating in this study and presented with an "Invitation to Participate in a Research Study" form ; the study assistant will obtain final consent if they agree. Those not interested in participating will simply receive their physician's standard bowel preparation protocol. There will be no coercion of any sort. Enrollment of participants will be performed with block randomizations of 2, 4, 6 and 8 by using a computer-generated table, with allocation concealment maintained through the use of consecutively numbered sealed envelopes. Colonoscopists and investigators will be blinded to allocation groups. Patients will be allocated to one of two groups: (1) Split dose Polyethylene Glycol Based Lavage (2L + 2L) with Standard dietary instructions- a low fibre diet for 4 days prior to colonoscopy and clear fluids after a low-fibre breakfast on the day before procedure; (2) Split dose Polyethylene Glycol Based Lavage (2L + 2L) with Low Fibre Lunch dietary instructions- a low fibre diet for 4 days prior to colonoscopy and clear fluids after a low-fibre breakfast and low-fibre lunch on the day before procedure

A study assistant will assign patients to their group based on the Randomization and instruct them on the proper use of their assigned bowel preparation method. Patients will be given a tolerability questionnaire, which has been modified from a previously used questionnaire, to be completed once their bowel preparation is finished and before coming to the CCSC for the colonoscopy (included in the appendix). Patient concerns or questions regarding the preparation will be directed toward the study assistant or clinic nurses as opposed to their endoscopist, so as to avoid un-blinding the Colonoscopist. The physician performing the procedure will then complete an Ottawa Bowel Preparation Scale, a validated Simplified Bowel Preparation scale and a New Bowel Prep Scale to assess colon cleanliness.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 to 74 Years referred to the Forzani & MacPhail Colon Cancer Screening Centre in Calgary, Alberta, Canada for Colonoscopy will be considered for inclusion.

Exclusion Criteria:

* Patients with acute Coronary Syndrome,
* Congestive Heart Failure,
* Unstable Angina,
* Known or suspected Renal Failure,
* Ascites,
* Known or suspected Bowel obstruction or
* Other comorbidities that may prevent Colonoscopy will be excluded.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 345 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-08 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Quality of Bowel Cleanliness | Procedure is completed (1 hour time). Questionnaires are manually entered by an assistant into the study database on the same day of collection.
  Ottawa bowel prep scale will be done by the Doctor to assess the quality of bowel cleanliness. The right, mid and rectosigmoid colon are each rated on a 5-point scale (0-4). Also a complete 3 point rating for overall colonic fluid is assessed giving an overall score range of 0-14. An excellent preperation should score 0-1, a good preparation 2-4, while scores >4 would indicate progressively worsening bowel preparations. A Simplified overall cleanliness score and a New bowel prep score will be completed and compared to the Ottawa scale.

SECONDARY OUTCOMES:
Patient satisfaction with preparation | Questionnaire given on the day of pre-screen will be collected on the day of colonoscopy, approximately 3 weeks. Patients are not followed or contacted past the day of colonoscopy.
  Patients will be given an anonymous tolerability questionnaire, which has been modified from a previously used questionnaire, to be completed once their bowel preparation is finished and before coming to the Centre for the Colonoscopy. The tool asks questions of patient satisfaction with preparation, ease or difficulty of completing the preparation and any side effects that have been experienced during the preparation.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Rostom, MD, Principal Investigator — University of Calgary
Locations (1):
- Forzani & MacPhail Colon Cancer Screening Centre, Alberta Health Services, Calgary, Alberta, Canada